CLINICAL TRIAL: NCT06331663
Title: To Explore the Optimal Dose of Remifentanil for Skull Pin Fixation Under Surgical Pleth Index Monitor in Intracranial Surgery
Brief Title: SPI and Remifentanil in Skull Pin Fixation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(II)-20240055
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-01

CONDITIONS: Pain, Procedural
Keywords: remifentanil, pain, surgical pleth index
MeSH Terms: conditions — Pain, Procedural; Pain | interventions — Remifentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): Neurosurgery with fixation
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — first start with remifentanil 5.0 ng/ml, and use the up and down method as adjust 0.5 ng/ml of concentration of remifentanil each time. Inadequate antinociception (Surgical Pleth Index(SPI) > 80 and hyperdynamics (the increased heart rate (HR) and mean blood pressure (MBP) above 20% of baseline or HR>100bpm and arterial blood pressure(ABP)>180/100mmHg)) is defined as failure, therefore we increase remifentanil by 0.5 ng/ml; otherwise, the setting is considered successful without abovementioned situations.

SUMMARY:
Forty patients were enrolled, and all patients used total intravenous anesthesia (remifentanil-propofol based total intravenous analgesia) as anesthesia induction and maintenance. According to the preliminary data of this department, patients who underwent intracranial surgery for skull pin fixation used remifentanil 5.0-6.0 ng/ml, while the hemodynamics is relatively stable. Therefore, when this plan is implemented, the patient needs to be under the same depth of anesthesia (monitored by electroencephalography, maintaining a value of 40-60), first start with remifentanil 5.0 ng/ml, and use the up and down method as adjust 0.5 ng/ml of concentration of remifentanil each time. Inadequate antinociception (Surgical Pleth Index(SPI) > 80 and hyperdynamics (the increased heart rate (HR) and mean blood pressure (MBP) above 20% of baseline or HR>100bpm and arterial blood pressure(ABP)>180/100mmHg)) is defined as failure, therefore we increase remifentanil by 0.5 ng/ml; otherwise, the setting is considered successful without abovementioned situations.

Data collection: heart rate, mean blood pressure, Surgical Pleth Index, bispectral Index, pulse pressure variance, systolic pressure variance, concentrations of propofol and remifentanil before 2 mins, during, 5, and 15 mins of skull pin fixation were recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 20 years old and less than 80 years old
2. With anesthesia risk grade below grade three (including grade three) (ASA I~III).
3. Patients who are expected to undergo intracranial surgery for skull pin fixation

Exclusion Criteria:

1. Those with anesthesia risk classification ASA class IV or higher
2. Those who are allergic to opioid analgesics or propofol drugs
3. Emergency patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
50% effect concentration of remifentanil | peri-fixation period
  50% effect concentration of remifentanil will be recorded at 2 mins before fixation, during fixation, 5 mins after fixation, and 15 mins after fixation.
90% effect concentration of remifentanil | peri-fixation period
  90% effect concentration of remifentanil will be recorded at 2 mins before fixation, during fixation, 5 mins after fixation, and 15 mins after fixation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan